CLINICAL TRIAL: NCT00992745
Title: A Phase I Pilot Study Comparing 123I MIP 1072 Versus 111In Capromab Pendetide in Subjects With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TX-P103
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; imaging; metastases; PSMA; ProstaScint®
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Capromab Pendetide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Previous ProstaScint® (Experimental): Subjects with a previous 111-In capromab pendetide image of sufficient quality obtained within 60 days of study enrollment will receive 123-I-MIP-1072 alone.
  Interventions: Drug: 123-I-MIP-1072
- No Previous ProstaScint® (Experimental): Subjects without a previous 111-In capromab pendetide image of sufficient quality obtained within 60 days of study enrollment will receive 123-I-MIP-1072 and 111-In capromab pendetide imaging.
  Interventions: Drug: 123-I-MIP-1072; Drug: 111-In capromab pendetide

INTERVENTIONS:
Drug: 123-I-MIP-1072 — Single 10 mCi intravenous injection
  Other Names: Trofex
Drug: 111-In capromab pendetide — Single 5 mCi intravenous injection
  Other Names: ProstaScint®
  Arms: No Previous ProstaScint®
Drug: 123-I-MIP-1072 — Single 5 mCi intravenous injection
  Other Names: Trofex

SUMMARY:
This is an open-label study comparing the imaging characteristics of 123-I-MIP-1072 and ProstaScint® (111-In-capromab pendetide)in patients with metastatic prostate cancer. Eligible patients will receive a dose of 123-I-MIP-1072 and have imaging studies and safety assessments (physical examination, vital signs, electrocardiogram, clinical laboratory tests) performed during the subsequent 24 hours. Two weeks later, patients will return for additional safety assessments and will receive ProstaScint® if they don't already have a pre-existing ProstaScint scan. Final assessments will be performed two weeks after the ProstaScint® scan unless there is a difference between the 123-I-MIP-1072 and ProstaScint® scans. If this is the case, another dose of 123-I-MIP-1072 will be given 12 weeks later, and imaging studies repeated.

ELIGIBILITY:
Subjects must meet all of the following criteria to be enrolled in this study.

1. Male aged 18 years or older
2. Signed written informed consent and willingness to comply with protocol requirements
3. Histologic diagnosis of prostate cancer by validated history and/or biopsy of the prostate or of a metastatic lesion.
4. Evidence of metastatic disease as documented by an abnormal bone scan and CT scan or MRI plus:

   * Castration/anti androgen therapy naïve/sensitive:

     1. Gleason Score ≥ 7 and PSA ≥ 2.0 ng/mL with history of prostatectomy or primary radiation therapy of the prostate gland and prior undetectable PSA or; PSA > 10.0 ng/mL if intact prostate, or
     2. Gleason score ≤ 6 and PSA is ≥ 20 ng/mL, or
     3. Gleason Score ≥ 8 and any doubling of PSA, or PSA > 0.5 ng/mL, or
     4. Clinical Stage 3 and Gleason Score ≥ 8

   If on anti androgen therapy, must have initiated therapy at least 4 weeks prior to treatment.
   * Castration/anti androgen therapy resistant:

     1. Patients must have current or historical evidence of disease progression concomitant with surgical (orchiectomy) or medical castration (LHRH analogue); anti androgen withdrawal (4 weeks for flutamide and 6 weeks for nilutamide or bicalutamide) is necessary only for patients on anti androgens who have demonstrated a > 3 month duration of beneficial response to anti androgens; progression is demonstrated by any of the following:

   I. PSA progression: 2 serial rising PSA determinations at least 14 days apart over the PSA nadir, with the last measurement ≥ 2 ng/mL

   II. Progression of measurable disease, or progression of non measurable disease as defined by:

   i. Soft tissue disease: The appearance of one or more new lesions, and/or unequivocal worsening of non measurable disease when compared to imaging studies acquired during castration therapy or against the precastration studies if there was no response, or ii. Bone disease: Appearance of two or more new areas of abnormal uptake on bone scan when compared to imaging studies acquired during castration therapy or against the pre castration studies if there was no response.

   III. Increased uptake of pre existing lesions on bone scan does not constitute progression.

   IV. Testosterone ≤ 50 ng/dL achieved via medical or surgical castration.
5. Male subjects who are fertile agree to use an acceptable form of birth control, defined as abstinence, barrier or other acceptable, effective contraceptive method throughout the study period. A second form of barrier birth control must be utilized if a subject's partner is using oral contraception until at least seven days after the last injection.
6. Karnofsky performance is ≥ 50
7. Adequate hematologic, renal and liver function:

   * WBC ≥ 2.0×103/mm3 (ANC > 1.0 x 103 mm3)
   * Platelet count ≥ 75×103/mm3
   * Hemoglobin ≥ 9.0 g/dL
   * Creatinine ≤ 2.5 mg/dL
   * Total bilirubin ≤ 2x ULN
   * AST, ALT ≤ 5x ULN

Exclusion Criteria:

1. Karnofsky performance status of < 50
2. Subject has received a permanent prostate brachytherapy implant within the last 3 months for 103Pd implants or 12 months for 125I implants
3. Subject was administered a diagnostic radioisotope within 5 physical half lives of that radioisotope prior to study enrollment
4. Subject has received an investigational compound and/or medical device or has been part of an investigational study within the past 30 days before enrollment into this study
5. Any treatment with radiopharmaceuticals, e.g. Strontium 89 and Samarium 153 within 6 months prior to enrollment
6. Ketoconazole or anti androgens (flutamide, nilutamide, bicalutamide) within 4 weeks prior to enrollment. Patients who demonstrate an antiandrogen withdrawal response, defined as a > 25% drop in PSA within 4 weeks (flutamide) or 6 weeks (nilutamide, bicalutamide) of stopping a non steroidal anti androgen, are not eligible until the PSA rises above the nadir observed after anti androgen withdrawal
7. Initiation of bisphosphonate therapy within 28 days prior to enrollment. Patients taking bisphosphonates should not have their dosing regimen altered unless medically warranted in the interval between baseline scans and end of study
8. Subject has any medical condition or other circumstances which, in the opinion of the Investigator, would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post dose follow up examinations
9. Subject is determined by the Investigator to be clinically unsuitable for the study
10. If the subject has had any other malignancies within the past year, other than basal or squamous cell carcinoma of the skin, diagnosis and location must be defined or be defined as clinically controlled or treated to complete response

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Estimate the imaging sensitivity and specificity of 10.0 mCi or 5.0 mCi of 123I MIP 1072 compared to 5 mCi of 111In capromab pendetide in subjects with metastatic prostate cancer by determining the presence and extent of the disease. | 24 hours post-injection

SECONDARY OUTCOMES:
Examine the imaging sensitivity and specificity of 10.0 mCi or 5.0 mCi of 123I MIP 1072 compared to 5 mCi of 111In capromab pendetide on a per lesion basis in subjects with metastatic prostate cancer | Through 2 weeks post-injection
To describe the safety of administering 10.0 mCi and 5.0 mCi of 123I MIP 1072 for the detection of metastatic prostate cancer | Through 2 weeks post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Dobkin, MD, Principal Investigator — Pacific Coast Imaging; Stanley Goldsmith, MD, Principal Investigator — NY Presbyterian Hospital - Weill Cornell Medical Center; Edward Coleman, MD, Principal Investigator — Duke University; Arif Hussain, MD, Principal Investigator — University of Maryland; Mack Roach, MD, Principal Investigator — University of California, San Francisco; Kevin Slawin, MD, Principal Investigator — Vanguard Urologic Research Foundation; Samuel L Kipper, MD, Principal Investigator — West Coast Radiology Centerse
Locations (7):
- United States (7):
  - West Coast Radiology Centers, Laguna Niguel, California
  - Pacific Coast Imaging, Newport Beach, California
  - University of California - San Francisco, San Francisco, California
  - University of Maryland, Baltimore, Maryland
  - New York Presbyterian Hospital - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vanguard Urologic Research Foundation, Houston, Texas